CLINICAL TRIAL: NCT02731170
Title: Effectiveness of Intensive Rehabilitation in Advanced Stages of Parkinson's Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Principal Investigator, Ilaria Zivi, MD, Ospedale Generale Di Zona Moriggia-Pelascini
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rehabilitation and PD
Record Dates: First submitted 2016-04-02; First posted 2016-04-07 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Advanced Stages; Rehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rehabilitation treatment (MIRT) (Experimental): MIRT consists of a 4-week physical therapy. daily sessions are subdivided in: motor treatment (2 hour), occupational therapy (1 hour) and speech Therapy (1 hour)
  Interventions: Behavioral: MIRT

INTERVENTIONS:
Behavioral: MIRT — MIRT consists of a 4-week physical therapy, in a hospital setting, which entails four daily sessions for five days and one hour of physical exercise on the sixth day. The duration of each session is about one hour. The first session consists of a one-to-one session with physical therapist involving muscle stretching. The second session includes aerobic exercises to improve balance and gait using different devices: a stabilometric platform, treadmill plus, crossover and cycloergometer. The third is a session of occupational therapy to improve autonomy in everyday activities. The last session includes one hour of speech therapy

SUMMARY:
this study is aimed to evaluate the effectiveness of an Multidisciplinary Intensive Rehabilitation Treatment in Advanced Stages of Parkinson's Disease.

In the last years, several evidences highlighted the need of a multidisciplinary and intensive approach to achieve good results in early stage of disease.

Hypothesis is that this approach is effectiveness also in moderate and advanced stages of disease

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a progressive neurodegenerative disease clinically characterized by motor and non-motor symptoms.

Dopamine replacement therapy (DRT) is the standard treatment for the motor symptom of PD, however DRT does not reduce axial PD symptoms such as freezing of gait, postural instability and balance disturbances. Further, long-term DRT could negatively impact on cognitive and motivational functions and leads to different motor and behavioural side effects. Therefore, the pharmacological approach becomes less effective in the moderate and advanced stages of disease.

The investigators testing the hypothesis that this approach is effectiveness also in moderate and advanced stages of disease In according with Hoehn and Yahr scale (H&Y) we identified 353 parkinsonian patients on stage 3, 79 subjects on stage 4 and 7 subjects on stage 5.

Clinical scores were assessed at baseline and after 4 weeks by neurologists and physiotherapists expert in movement disorders. All evaluations were performed in the morning, one hour after taking drugs. The assessment included: Unified Parkinson's Disease Rating Scale (UPDRS), for clinical evaluation, Berg Balance Scale (BBS), Timed Up and Go Test (TUG), Six Minutes Walking Test (6MWT), Freezing of Gait Questionnaire (FOGQ) and Abnormal Involuntary Movements Scale (AIMS) for motor symptoms evaluation and, finally, Parkinson's Disease Disability Scale (PDDS), for evaluation of the functional impact of the disease. Since in the advanced stages of PD one of the most troublesome complication includes cognitive disorders, a Neuropsychologist performed a cognitive assessment at the admission. The neuropsychological profile was explored using the Mini Mental State Examination (MMSE), a tool for screening of cognitive impairment, and the Frontal Assessment Battery (FAB) for the evaluation of frontal lobe dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

clinica diagnosis of Parkinson Disease

Exclusion Criteria:

comorbidity with other neurological conditions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 439 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson Disease Rating Scale | 4 weeks
six-minutes walking test | 4 weeks
Time up and go Test | 4 weeks
Berg Balance Scale | 4 weeks
Freezing of Gait Questionnaire | 4 weeks
Parkinson's Disease Disability Scale | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Parkinson's Disease and Brain Injury Rehabilitation, of the 'Moriggia-Pelascini' Hospital, Gravedona Ed Uniti, Como, Italy

IPD SHARING:
Plan to Share IPD: No